CLINICAL TRIAL: NCT01976741
Title: An Open Label, Non-randomized, Phase I Dose Escalation Study to Characterize Safety, Tolerability, Pharmacokinetics and Maximum Tolerated Dose of BAY1163877 in Subjects With Refractory, Locally Advanced or Metastatic Solid Tumors
Brief Title: Dose Escalation Pan-FGFR (Fibroblast Growth Factor Receptor) Inhibitor (Rogaratinib)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16443; 2013-002155-15 (EudraCT Number)
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Neoplasms
Keywords: Phase I; Dose escalation; refractory, locally advanced or metastatic solid tumor; Bladder cancer; squamous non-small cell lung cancer; pan-FGFR inhibitor; lung adenocarcinoma; head and neck cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Urinary Bladder Neoplasms; Adenocarcinoma of Lung; Head and Neck Neoplasms | interventions — Rogaratinib; Solutions; Tablets; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Rogaratinib total dose escalation (Experimental): Participants with any type of solid tumor received escalating doses of Rogaratinib oral solution or tablet. The actual dose-escalation cohorts were 100 mg (50 mg BID), 200 mg (100 mg BID), 400 mg (200 mg BID), 800 mg (400 mg BID), 1200 mg (600 mg BID), and 1600 mg (800 mg BID). The participants in the 100 mg and 200 mg dose-escalation cohorts received oral solution and the participants in all the subsequent dose-escalation cohorts received tablet. And as an exception, on C1D-3 in the 200 mg dose-escalation cohort, the participants received tablet instead of oral solution.
  Interventions: Drug: Rogaratinib (BAY1163877) oral solution; Drug: Rogaratinib (BAY1163877) oral tablet
- Rogaratinib dose expansion (All Comers) (Experimental): Participants with cancer types other than bladder cancer (BC), squamous cell carcinoma of the head and neck (SCCHN), and squamous non-small cell lung cancer (sqNSCLC) received 800 mg Rogaratinib oral tablet b.i.d.
  (1600 mg/day) in 21-days cycles.
  Interventions: Drug: Rogaratinib (BAY1163877) 800 mg BID
- Rogaratinib dose expansion (BC) (Experimental): Participants with bladder cancer (BC) received 800 mg Rogaratinib oral tablet b.i.d. (1600 mg/day) in 21-days cycles.
  Interventions: Drug: Rogaratinib (BAY1163877) 800 mg BID
- Rogaratinib dose expansion (SCCHN) (Experimental): Participants with squamous cell carcinoma of the head and neck (SCCHN) received 800 mg Rogaratinib oral tablet b.i.d. (1600 mg/day) in 21-days cycles.
  Interventions: Drug: Rogaratinib (BAY1163877) 800 mg BID
- Rogaratinib dose expansion (sqNSCLC) (Experimental): Participants with squamous non-small cell lung cancer (sqNSCLC) received 800 mg Rogaratinib oral tablet b.i.d. (1600 mg/day) in 21-days cycles.
  Interventions: Drug: Rogaratinib (BAY1163877) 800 mg BID

INTERVENTIONS:
Drug: Rogaratinib (BAY1163877) oral solution — Participants received Rogaratinib oral solution as a single dose on Cycle 1 Day 1 (C1D1) and twice daily (BID) from Cycle 1 Day 3 (C1D3) onward for the remaining 19 days of Cycle 1. For subsequent cycles, study drug was administered twice daily for 21 days each Cycle.
  Arms: Rogaratinib total dose escalation
Drug: Rogaratinib (BAY1163877) oral tablet — Participants received Rogaratinib oral tablet as a single dose on C1D1 and BID from C1D3 onward for the remaining 19 days of Cycle 1. For subsequent cycles, study drug was administered twice daily for 21 days each Cycle.
  Arms: Rogaratinib total dose escalation
Drug: Rogaratinib (BAY1163877) 800 mg BID — Participants received Rogaratinib 800 mg oral tablet as a single dose on C1D1 and BID (in total 1600 mg) from C1D3 onward for the remaining 19 days of Cycle 1. For subsequent cycles, study drug was administered twice daily for 21 days each Cycle.
  Arms: Rogaratinib dose expansion (All Comers); Rogaratinib dose expansion (BC); Rogaratinib dose expansion (SCCHN); Rogaratinib dose expansion (sqNSCLC)

SUMMARY:
* This was the first study where BAY1163877 was given to humans. Impact of the study was to evaluate if patients with advanced solid cancers show advanced clinical benefit under the treatment with the pan FGFR inhibitor. Patients (all comers) received the study drug treatment in a dose-escalation scheme (no placebo group) to determine the safety, tolerability and maximum tolerated dose (MTD) of BAY1163877. The relative bioavailability of liquid service formulation and tablets was determined.
* After the MTD was defined patients with solid tumors (all comers), lung cancer (lung adenocarcinoma & squamous non-small cell lung cancer), head and neck cancer or bladder cancer was enrolled according to their FGFR expression profile (biomarker stratification).
* The study also assessed the pharmacokinetics, biomarker status, pharmacodynamic parameters and tumor response of BAY1163877.
* BAY1163877 was given twice daily as oral application. Treatment was stopped if the tumor continued to grow, if side effects, which the patient cannot tolerate, occurred or if the patient decided to exit treatment.

ELIGIBILITY:
Inclusion Criteria:

* For dose escalation: Participants with any type of solid tumor (all comer) were eligible for dose escalation and dose expansion at MTD in Part 1; Participants enrolled for dose expansion (MTD expansion cohort "all comer") were stratified according to high fibroblast growth factor receptor (FGFR) expression levels / FGFR mutation using archival or fresh tumor biopsy material
* For expansion cohorts: Participants were eligible for Part 2 only if they have histological or cytological confirmed squamous non-small cell lung cancer (sqNSCLC), lung adenocarcinoma, head and neck cancer or bladder cancer (BC). All participants in Part 2 were stratified according to high FGFR expression levels FGFR mutation using archival or fresh tumor biopsy specimen. BC participants with low overall FGFR expression levels could be included if activating FGFR3 (FGFR tyrosine kinases 3) mutations were confirmed
* Participants must have measurable disease (Response evaluation criteria in solid tumors (RECIST 1.1))
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2
* Bone marrow, liver and renal functions as assessed by adequate laboratory methods to be conducted within 7 days prior to starting study Treatment
* Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m^2 according to the modified diet in renal disease (MDRD) abbreviated formula

Exclusion Criteria:

* Previous treatment with anti-FGFR directed therapies (e.g. receptor tyrosine kinase inhibitors or FGFR-specific antibodies)
* Concomitant therapies that cannot be discontinued or switched to a different medication prior to study entry that are known to increase serum phosphate levels are not permitted within 4 weeks prior to start of study treatment)
* Anticancer chemotherapy or immunotherapy during the study or within 5-halflives prior to start of study treatment. Mitomycin C, nitrosoureas or monoclonal antibodies with anticancer activity (e.g. bevacizumab or cetuximab etc.) should not be given within 6 weeks before starting to receive study treatment or within 6 weeks of pre-treatment biopsy for biomarker (p-ERK1/2) studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2013-12-30 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (24):
- United States (2):
  - Chicago, Illinois
  - Pittsburgh, Pennsylvania
- France (5):
  - Besançon
  - Créteil
  - Dijon
  - Lille
  - Lyon
- Germany (9):
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Weiden, Bavaria
  - Würzburg, Bavaria
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Dresden, Saxony
  - Hamburg
  - Magdeburg
- Singapore, Singapore
- Seoul, South Korea
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia
- Switzerland (3):
  - Sankt Gallen, Canton of St. Gallen
  - Chur, Kanton Graubünden
  - Geneva

REFERENCES:
- [Result] Schuler M, Cho BC, Sayehli CM, Navarro A, Soo RA, Richly H, Cassier PA, Tai D, Penel N, Nogova L, Park SH, Schostak M, Gajate P, Cathomas R, Rajagopalan P, Grevel J, Bender S, Boix O, Nogai H, Ocker M, Ellinghaus P, Joerger M. Rogaratinib in patients with advanced cancers selected by FGFR mRNA expression: a phase 1 dose-escalation and dose-expansion study. Lancet Oncol. 2019 Oct;20(10):1454-1466. doi: 10.1016/S1470-2045(19)30412-7. Epub 2019 Aug 9. PMID 31405822
- [Result] Grunewald S, Politz O, Bender S, Heroult M, Lustig K, Thuss U, Kneip C, Kopitz C, Zopf D, Collin MP, Boemer U, Ince S, Ellinghaus P, Mumberg D, Hess-Stumpp H, Ziegelbauer K. Rogaratinib: A potent and selective pan-FGFR inhibitor with broad antitumor activity in FGFR-overexpressing preclinical cancer models. Int J Cancer. 2019 Sep 1;145(5):1346-1357. doi: 10.1002/ijc.32224. Epub 2019 Mar 13. PMID 30807645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 29 centers in 7 countries, between 30 Dec 2013 (first subject first visit) and 27 Nov 2019 (last subject last visit).
Pre-assignment Details: A total of 988 participants were screened, of whom 168 participants were assigned into the study and received at least one dose of study medication.
Groups:
- Rogaratinib 50 mg BID: Participants received Rogaratinib as a single dose of 50 mg solution on C1D1 and 50 mg solution BID (in total 100 mg) from C1D3 ongoing in 21-days cycles in dose escalation phase.
- Rogaratinib 100 mg BID: Participants received a single dose of 100 mg Rogaratinib tablet formulation on C1D-3, followed by a single dose of 100 mg solution on C1D1 and continued with 100 mg BID of solution (in total 200 mg) from C1D3 ongoing in 21-days cycles in dose escalation phase.
- Rogaratinib 200 mg BID: Participants received Rogaratinib as a single dose of 200 mg tablet on C1D1 and 200 mg tablet BID (in total 400 mg) from C1D3 ongoing in 21-days cycles in dose escalation phase.
- Rogaratinib 400 mg BID: Participants received Rogaratinib as a single dose of 400 mg tablet on C1D1 and 400 mg tablet BID (in total 800 mg) from C1D3 ongoing in 21-days cycles in dose escalation phase.
- Rogaratinib 600 mg BID: Participants received Rogaratinib as a single dose of 600 mg tablet on C1D1 and 600 mg tablet BID (in total 1200 mg) from C1D3 ongoing in 21-days cycles in dose escalation phase.
- Rogaratinib 800 mg BID: Participants received Rogaratinib as a single dose of 800 mg tablet on C1D1 and 800 mg tablet BID (in total 1600 mg) from C1D3 ongoing in 21-days cycles in dose escalation phase.
- Rogaratinib Dose Expansion (All Comers): Participants with cancer types other than bladder cancer (BC), squamous cell carcinoma of the head and neck (SCCHN), and squamous non-small cell lung cancer (sqNSCLC) received 800 mg Rogaratinib oral tablet BID (1600 mg/day) in 21-days cycles.
- Rogaratinib Dose Expansion (BC): Participants with bladder cancer (BC) received 800 mg Rogaratinib oral tablet BID (1600 mg/day) in 21-days cycles.
- Rogaratinib Dose Expansion (SCCHN): Participants with squamous cell carcinoma of the head and neck (SCCHN) received 800 mg Rogaratinib oral tablet BID (1600 mg/day) in 21-days cycles.
- Rogaratinib Dose Expansion (sqNSCLC): Participants with squamous non-small cell lung cancer (sqNSCLC) received 800 mg Rogaratinib oral tablet BID (1600 mg/day) in 21-days cycles.
Period: Overall Study
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Started | 4 | 4 | 4 | 3 | 4 | 4 | 23 | 74 | 8 | 40
Completed | 3 | 4 | 1 | 2 | 4 | 4 | 19 | 62 | 7 | 36
Not Completed | 1 | 0 | 3 | 1 | 0 | 0 | 4 | 12 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 8 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC) | Total
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 4 | 23 | 74 | 8 | 40 | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (20.4) | 58.5 (12.4) | 55.8 (15.3) | 56.3 (9.8) | 56.8 (12.9) | 64.3 (8.4) | 63.0 (7.8) | 66.4 (8.6) | 63.4 (11.1) | 62.6 (6.6) | 63.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 1 | 1 | 0 | 9 | 20 | 0 | 8 | 46
  Male | 1 | 2 | 2 | 2 | 3 | 4 | 14 | 54 | 8 | 32 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 4 | 3 | 4 | 4 | 23 | 61 | 8 | 34 | 149
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 1 | 1 | 8 | 13 | 1 | 11 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 4 | 3 | 2 | 3 | 3 | 15 | 50 | 7 | 22 | 113
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 7 | 18
Eastern Cooperative Oncology Group (ECOG) Performance status [Count of Participants; unit: Participants] — ECOG score: 0=fully active; 1=restricted active; 2=ambulatory and capable of all self-care.
  Participants
    ECOG=0 | 2 | 1 | 1 | 1 | 2 | 2 | 10 | 20 | 3 | 14 | 56
    ECOG=1 | 2 | 3 | 3 | 2 | 1 | 1 | 12 | 49 | 5 | 22 | 100
    ECOG=2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 5 | 0 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD), Defined as Maximum Dose at Which the Incidence of Dose Limiting Toxicities (DLTs) During Cycle 1 is Below 20%
Description: The MTD was defined as maximum dose at which the incidence of Dose Limiting Toxicities (DLTs) during Cycle 1 is below 20%. DLT was defined as any of the pre-defined adverse events occurring during Cycle 1 of a dose level and regarded by the investigators and/or sponsor to be related to the investigational drug. BID=twice daily.
Time Frame: Up to 21 days
Population: MTD evaluation set: All participants of the total dose-escalation group who completed Cycle 1 or discontinued during Cycle 1 due to an adverse event or DLT.
Measure: Number; unit: mg BID
Arm/Group | Rogaratinib Total Dose Escalation
Number analyzed (Participants) | 21
mg BID | 800

2. Primary Outcome: Number of DLTs During Cycle 1
Description: DLT was defined as any of the pre-defined adverse events occurring during Cycle 1 of a dose level and regarded by the investigators and/or sponsor to be related to the investigational drug.
Time Frame: Up to 21 days
Population: as for outcome 1
Measure: Number; unit: DLTs
Arm/Group | Rogaratinib Total Dose Escalation
Number analyzed (Participants) | 21
DLTs | 0

3. Primary Outcome: Cmax (Maximum Drug Concentration in Plasma) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3
Description: Maximum drug concentration in plasma (Cmax) of BAY1163877 after single dose administration on Cycle 1, Day -3. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day -2) and 48 hour(s) post-dose (Day -1)
Population: All participants with valid pharmacokinetic (PK) data on Cycle 1, Day -3. Some of the participants from the expansion cohorts were included in Rogaratinib expansion food effect.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Groups:
- Rogaratinib Expansion Food Effect: For food effect assessment, participants in the MTD expansion cohorts (1600 mg) of study Part 1 and Part 2 received single doses (800 mg) of the study drug on C1D-3 (after consumption of a high-fat, high-calorie breakfast) and on C1D1 (after an overnight fast of at least 8 h). The participants continued with 800 mg BID doses of the study drug from C1D3 onward.
Arm/Group | Rogaratinib 100 mg BID | Rogaratinib Expansion Food Effect
Number analyzed (Participants) | 4 | 10
µg/L | 2760 (56.5) | 11300 (33.8)

4. Primary Outcome: Cmax (Maximum Drug Concentration in Plasma) of BAY1163877 After Single Dose Administration on Cycle 1, Day 1
Description: Maximum drug concentration in plasma (Cmax) of BAY1163877 after single dose administration on Cycle 1, Day 1. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day 1) and 48 hour(s) post-dose (Day 2)
Population: All participants with valid PK data on Cycle 1, Day 1. Some of the participants from the expansion cohorts were included in Rogaratinib expansion food effect, and participants who received 800 mg BID in either escalation or expansion phase were combined as pre-specified in the Statistical Analysis Plan.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Groups:
- Rogaratinib 800 mg BID Pooled: Participants received Rogaratinib 800 mg tablet BID (in total 1600 mg) in dose escalation phase and MTD expansion phase.
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 4 | 3 | 4 | 4 | 51 | 11 | 19 | 13 | 2 | 13
µg/L | 3640 (16.8) | 4360 (36.4) | 5630 (46.2) | 9480 (16.1) | 9060 (32.3) | 10200 (17.3) | 11000 (34.3) | 11000 (47.6) | 10900 (32.5) | 11000 (48.1) | 13900 (52.6) | 11200 (26.0)

5. Primary Outcome: AUC(0-12) (Area Under the Plasma Concentration vs Time Curve From Time Zero to 12 Hours) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3
Description: Area under the plasma concentration vs time curve from time zero to 12 hours (AUC(0-12)) of BAY1163877 after single dose administration on Cycle 1, Day -3. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day -2) and 48 hour(s) post-dose (Day -1)
Population: All participants with valid PK data on Cycle 1, Day -3. Some of the participants from the expansion cohorts were included in Rogaratinib expansion food effect.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/L
Arm/Group | Rogaratinib 100 mg BID | Rogaratinib Expansion Food Effect
Number analyzed (Participants) | 4 | 10
µg*h/L | 15600 (72.0) | 71000 (42.7)

6. Primary Outcome: AUC(0-12) (Area Under the Plasma Concentration vs Time Curve From Time Zero to 12 Hours) of BAY1163877 After Single Dose Administration on Cycle 1, Day 1
Description: Area under the plasma concentration vs time curve from time zero to 12 hours (AUC(0-12)) of BAY1163877 after single dose administration on Cycle 1, Day 1. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day 1) and 48 hour(s) post-dose (Day 2)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 4 | 4 | 51 | 11 | 19 | 13 | 2 | 13
µg*h/L | 12100 (16.3) | 15300 (41.4) | 33200 (33.1) | 44000 (68.9) | 54300 (31.3) | 55700 (43.5) | 63900 (45.0) | 74200 (49.7) | 63700 (46.5) | 59700 (56.4) | 101000 (37.4) | 66700 (32.0)

7. Primary Outcome: AUC(0-tlast) (Area Under the Plasma Concentration vs Time Curve From Time Zero to the Last Data Point > LLOQ [Lower Limit of Quantification]) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3
Description: Area under the plasma concentration vs time curve from time zero to the last data point > LLOQ [lower limit of quantification] (AUC(0-tlast)) of BAY1163877 after single dose administration on Cycle 1, Day -3. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day -2) and 48 hour(s) post-dose (Day -1)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/L
Arm/Group | Rogaratinib 100 mg BID | Rogaratinib Expansion Food Effect
Number analyzed (Participants) | 4 | 10
µg*h/L | 20000 (87.3) | 99300 (52.9)

8. Primary Outcome: AUC(0-tlast) (Area Under the Plasma Concentration vs Time Curve From Time Zero to the Last Data Point > LLOQ [Lower Limit of Quantification]) of BAY1163877 After Single Dose Administration on Cycle 1, Day 1
Description: Area under the plasma concentration vs time curve from time zero to the last data point > LLOQ [lower limit of quantification] (AUC(0-tlast)) of BAY1163877 after single dose administration on Cycle 1, Day 1. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day 1) and 48 hour(s) post-dose (Day 2)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 4 | 4 | 49 | 10 | 19 | 11 | 2 | 13
µg*h/L | 14200 (24.4) | 20100 (57.7) | 43800 (36.3) | 62000 (114) | 78000 (38.5) | 86600 (41.2) | 103000 (53.5) | 121000 (49.3) | 104000 (73.4) | 108000 (33.8) | 172000 (55.3) | 94900 (39.6)

9. Primary Outcome: AUC (Area Under the Plasma Concentration vs Time Curve From Zero to Infinity) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3
Description: Area under the plasma concentration vs time curve from zero to infinity (AUC) of BAY1163877 after single dose administration on Cycle 1, Day -3. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day -2) and 48 hour(s) post-dose (Day -1)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/L
Arm/Group | Rogaratinib 100 mg BID | Rogaratinib Expansion Food Effect
Number analyzed (Participants) | 4 | 10
µg*h/L | 20200 (87.1) | 102000 (55.2)

10. Primary Outcome: AUC (Area Under the Plasma Concentration vs Time Curve From Zero to Infinity) of BAY1163877 After Single Dose Administration on Cycle 1, Day 1
Description: Area under the plasma concentration vs time curve from zero to infinity (AUC) of BAY1163877 after single dose administration on Cycle 1, Day 1. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day 1) and 48 hour(s) post-dose (Day 2)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 4 | 3 | 46 | 10 | 18 | 11 | 2 | 12
µg*h/L | 14300 (24.5) | 20700 (58.1) | 44300 (37.1) | 64000 (118) | 79800 (39.5) | 95400 (48.7) | 109000 (58.4) | 133000 (53.3) | 109000 (77.5) | 115000 (38.9) | 191000 (69.9) | 99600 (46.5)

11. Primary Outcome: Cmax/D (Maximum Drug Concentration in Plasma Divided by Dose) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3
Description: Maximum drug concentration in plasma divided by dose (Cmax/D) of BAY1163877 after single dose administration on Cycle 1, Day -3. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day -2) and 48 hour(s) post-dose (Day -1)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /L
Arm/Group | Rogaratinib 100 mg BID | Rogaratinib Expansion Food Effect
Number analyzed (Participants) | 4 | 10
/L | 0.0276 (56.5) | 0.0141 (33.8)

12. Primary Outcome: Cmax/D (Maximum Drug Concentration in Plasma Divided by Dose) of BAY1163877 After Single Dose Administration on Cycle 1, Day 1
Description: Maximum drug concentration in plasma divided by dose (Cmax/D) of BAY1163877 after single dose administration on Cycle 1, Day 1. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day 1) and 48 hour(s) post-dose (Day 2)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 4 | 3 | 4 | 4 | 51 | 11 | 19 | 13 | 2 | 13
/L | 0.0728 (16.8) | 0.0436 (36.4) | 0.0282 (46.2) | 0.0237 (16.1) | 0.0151 (32.3) | 0.0127 (17.3) | 0.0138 (34.3) | 0.0137 (47.6) | 0.0137 (32.5) | 0.0137 (48.1) | 0.0174 (52.6) | 0.0140 (26.0)

13. Primary Outcome: AUC(0-12)/D (Area Under the Plasma Concentration vs Time Curve From Time Zero to 12 Hours Divided by Dose) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3
Description: Area under the plasma concentration vs time curve from time zero to 12 hours divided by dose (AUC(0-12)/D) of BAY1163877 after single dose administration on Cycle 1, Day -3. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day -2) and 48 hour(s) post-dose (Day -1)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h/L
Arm/Group | Rogaratinib 100 mg BID | Rogaratinib Expansion Food Effect
Number analyzed (Participants) | 4 | 10
h/L | 0.156 (72.0) | 0.0888 (42.7)

14. Primary Outcome: AUC(0-12)/D (Area Under the Plasma Concentration vs Time Curve From Time Zero to 12 Hours Divided by Dose) of BAY1163877 After Single Dose Administration on Cycle 1, Day 1
Description: Area under the plasma concentration vs time curve from time zero to 12 hours divided by dose (AUC(0-12)/D) of BAY1163877 after single dose administration on Cycle 1, Day 1. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day 1) and 48 hour(s) post-dose (Day 2)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h/L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 4 | 4 | 51 | 11 | 19 | 13 | 2 | 13
h/L | 0.242 (16.3) | 0.153 (41.4) | 0.166 (33.1) | 0.110 (68.9) | 0.0906 (31.1) | 0.0696 (43.5) | 0.0798 (45.0) | 0.0927 (49.7) | 0.0796 (46.5) | 0.0747 (56.4) | 0.126 (37.4) | 0.0834 (32.0)

15. Primary Outcome: AUC(0-tlast)/D (Area Under the Plasma Concentration vs Time Curve From Time Zero to the Last Data Point > LLOQ Divided by Dose) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3
Description: Area under the plasma concentration vs time curve from time zero to the last data point > LLOQ divided by dose (AUC(0-tlast)/D) of BAY1163877 after single dose administration on Cycle 1, Day -3. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day -2) and 48 hour(s) post-dose (Day -1)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h/L
Arm/Group | Rogaratinib 100 mg BID | Rogaratinib Expansion Food Effect
Number analyzed (Participants) | 4 | 10
h/L | 0.200 (87.3) | 0.124 (52.9)

16. Primary Outcome: AUC(0-tlast)/D (Area Under the Plasma Concentration vs Time Curve From Time Zero to the Last Data Point > LLOQ Divided by Dose) of BAY1163877 After Single Dose Administration on Cycle 1, Day 1
Description: Area under the plasma concentration vs time curve from time zero to the last data point > LLOQ divided by dose (AUC(0-tlast)/D) of BAY1163877 after single dose administration on Cycle 1, Day 1. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day 1) and 48 hour(s) post-dose (Day 2)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h/L
Groups:
- Rogaratinib Dose Expansion (All Comers): Participants with cancer types other than bladder cancer (BC), squamous cell carcinoma of the head and neck (SCCHN), and squamous non-small cell lung cancer (sqNSCLC) received 800 mg Rogaratinib oral tablet BID (1600 mg/day) in 21- days cycles.
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 4 | 4 | 49 | 10 | 19 | 11 | 2 | 13
h/L | 0.283 (24.4) | 0.201 (57.7) | 0.219 (36.3) | 0.155 (114) | 0.130 (38.5) | 0.108 (41.2) | 0.129 (53.5) | 0.152 (49.3) | 0.130 (73.4) | 0.135 (33.8) | 0.215 (55.3) | 0.119 (39.6)

17. Primary Outcome: AUC/D (AUC Divided by Dose) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3
Description: AUC divided by dose (AUC/D) of BAY1163877 after single dose administration on Cycle 1, Day -3. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day -2) and 48 hour(s) post-dose (Day -1)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h/L
Arm/Group | Rogaratinib 100 mg BID | Rogaratinib Expansion Food Effect
Number analyzed (Participants) | 4 | 10
h/L | 0.202 (87.1) | 0.127 (55.2)

18. Primary Outcome: AUC/D (AUC Divided by Dose) of BAY1163877 After Single Dose Administration on Cycle 1, Day 1
Description: AUC divided by dose (AUC/D) of BAY1163877 after single dose administration on Cycle 1, Day 1. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (Day 1) and 48 hour(s) post-dose (Day 2)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h/L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 4 | 3 | 46 | 10 | 18 | 11 | 2 | 12
h/L | 0.286 (24.5) | 0.207 (58.1) | 0.221 (37.1) | 0.160 (118) | 0.133 (39.5) | 0.119 (48.7) | 0.137 (58.4) | 0.166 (53.3) | 0.136 (77.5) | 0.144 (38.9) | 0.239 (69.9) | 0.124 (46.5)

19. Primary Outcome: Cmax,md (Cmax After Multiple-dose Administration) of BAY1163877 on Cycle 1, Day 15
Description: Cmax,md (Cmax after multiple-dose administration) of BAY1163877. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose (before morning dose), and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
Population: All participants with valid PK data on Cycle 1, Day 15. Some of the participants from the expansion cohorts were included in Rogaratinib expansion food effect, and participants who received 800 mg BID in either escalation or expansion phase were combined as pre-specified in the Statistical Analysis Plan.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 4 | 70 | 7 | 15 | 27 | 1 | 23
µg/L | 3940 (38.5) | 4870 (35.2) | 8320 (68.9) | 9490 (63.1) | 10500 (32.6) | 12400 (33.8) | 12600 (34.6) | 11000 (27.9) | 12300 (31.0) | 13100 (33.6) | 13100 | 12300 (40.5)

20. Primary Outcome: Cmax/Dmd (Cmax Divided by Dose After Multiple-dose Administration) of BAY1163877 on Cycle 1, Day 15
Description: Cmax/Dmd (Cmax divided by dose after multiple-dose administration) of BAY1163877. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose (before morning dose), and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 4 | 70 | 7 | 15 | 27 | 1 | 23
/L | 0.0789 (38.5) | 0.0487 (35.2) | 0.0416 (68.9) | 0.0237 (63.1) | 0.0174 (32.6) | 0.0155 (33.8) | 0.0158 (34.6) | 0.0138 (27.9) | 0.0154 (31.0) | 0.0163 (33.6) | 0.0163 | 0.0153 (40.5)

21. Primary Outcome: AUC(0-12)md (AUC(0-12) After Multiple-dose Administration) of BAY1163877 on Cycle 1, Day 15
Description: AUC(0-12)md (AUC(0-12) after multiple-dose administration) of BAY1163877. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose (before morning dose), and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 4 | 69 | 7 | 15 | 27 | 1 | 22
µg*h/L | 13300 (75.4) | 21500 (98.5) | 41700 (27.9) | 61100 (66.2) | 73500 (33.4) | 90900 (28.8) | 85300 (42.8) | 87100 (28.5) | 81700 (44.5) | 84500 (40.8) | 106000 | 87100 (49.1)

22. Primary Outcome: AUC(0-12)/Dmd (AUC(0-12) Divided by Dose After Multiple-dose Administration) of BAY1163877 on Cycle 1, Day 15
Description: AUC(0-12)/Dmd (AUC(0-12) divided by dose after multiple-dose administration) of BAY1163877. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose (before morning dose), and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h/L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 4 | 69 | 7 | 15 | 27 | 1 | 22
h/L | 0.266 (75.4) | 0.215 (98.5) | 0.209 (27.9) | 0.153 (66.2) | 0.123 (33.4) | 0.114 (28.8) | 0.107 (42.8) | 0.109 (28.5) | 0.102 (44.5) | 0.106 (40.8) | 0.132 | 0.109 (49.1)

23. Primary Outcome: AUC(0-tlast)md (AUC(0-tlast) After Multiple Dose Administration) of BAY1163877 on Cycle 1, Day 15
Description: AUC(0-tlast)md (AUC(0-tlast) after multiple dose administration) of BAY1163877. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose (before morning dose), and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 4 | 70 | 7 | 15 | 27 | 1 | 23
µg*h/L | 12500 (78.5) | 21500 (99.8) | 39200 (19.1) | 60200 (65.8) | 72500 (33.3) | 89000 (30.9) | 81500 (43.4) | 84100 (31.3) | 75000 (44.3) | 83600 (40.8) | 103000 | 81300 (50.1)

24. Primary Outcome: AUC(0-tlast)/Dmd (AUC(0-tlast) Divided by Dose After Multiple-dose Administration) of BAY1163877 on Cycle 1, Day 15
Description: AUC(0-tlast)/Dmd (AUC(0-tlast) divided by dose after multiple-dose administration) of BAY1163877. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose (before morning dose), and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h/L
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 4 | 70 | 7 | 15 | 27 | 1 | 23
h/L | 0.250 (78.5) | 0.215 (99.8) | 0.196 (19.1) | 0.151 (65.8) | 0.121 (33.3) | 0.111 (30.9) | 0.102 (43.4) | 0.105 (31.3) | 0.0937 (44.3) | 0.105 (40.8) | 0.129 | 0.102 (50.1)

25. Primary Outcome: %AE,ur(0-12) (Amount of Drug Excreted Via Urine During the Collection Interval 0 - 12 Hours Post Administration) of BAY1163877
Description: %AE,ur(0-12) (amount of drug excreted via urine during the collection interval 0 - 12 hours post administration, also expressed as percent of dose administered) of BAY1163877.
Time Frame: On Cycle1, Day 1
Population: Urine interval samples on C1D1 were collected in a subgroup of subjects from the 800 mg BID expansion part.
Measure: Median (Full Range); unit: percentage
Arm/Group | Rogaratinib 800 mg BID Pooled
Number analyzed (Participants) | 13
percentage | 0.164 [0.0363 to 0.665]

26. Primary Outcome: %AE,ur(0-24) (Amount of Drug Excreted Via Urine During the Collection Interval 0 - 24 Hours Post Administration) of BAY1163877
Description: %AE,ur(0-24) (amount of drug excreted via urine during the collection interval 0 - 24 hours post administration, also expressed as percent of dose administered) of BAY1163877.
Time Frame: On Cycle1, Day 1
Population: Urine interval samples on C1D1 were collected in a subgroup of subjects from the 800 mg BID expansion part.
Measure: Median (Full Range); unit: percentage
Arm/Group | Rogaratinib 800 mg BID Pooled
Number analyzed (Participants) | 13
percentage | 0.180 [0.0587 to 0.695]

27. Primary Outcome: %AE,ur(12-24) (Amount of Drug Excreted Via Urine During the Collection Interval 12 - 24 Hours Post Administration) of BAY1163877
Description: %AE,ur(12-24) (amount of drug excreted via urine during the collection interval 12 - 24 hours post administration, also expressed as percent of dose administered) of BAY1163877.
Time Frame: On Cycle1, Day 1
Population: Urine interval samples on C1D1 were collected in a subgroup of subjects from the 800 mg BID expansion part.
Measure: Median (Full Range); unit: percentage
Arm/Group | Rogaratinib 800 mg BID Pooled
Number analyzed (Participants) | 13
percentage | 0.0224 [0.0107 to 0.0596]

28. Secondary Outcome: Response Rate as Defined by RECIST Version 1.1 Reported as Number of Participants With Different Response Type
Description: Response as defined by RECIST (Response Evaluation Criteria in Solid Tumors) version 1.1: complete response (CR: disappearance of all target lesions), partial response (PR: at least a 30% decrease in the sum of diameters of target lesions taking as the reference the baseline sum of diameters), stable disease (SD: steady state of disease. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as a reference, the smallest sum of diameters while in the trial), progressive disease (PD: at least a 20% increase in the sum of diameters of the target lesions, taking as a references the smallest sum on study).
Time Frame: Up to 2 years
Population: Participants received at least one dose of Rogaratinib and have post-baseline efficacy data available. Participants were grouped as described in the SAP to allow a comparison of all dose escalation patients (all dose levels pooled together), dose expansion patients (four groups) and total number of patients (overview summaries) in the same table.
Measure: Count of Participants; unit: Participants
Arm/Group | Rogaratinib Total Dose Escalation | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 21 | 22 | 70 | 7 | 37
Participants
  missing | 2 | 1 | 1 | 1 | 2
  CR | 0 | 0 | 1 | 0 | 0
  PD | 9 | 8 | 20 | 3 | 11
  PR | 0 | 1 | 14 | 1 | 2
  SD | 10 | 12 | 34 | 2 | 22

29. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time (days) from the date of the first dose of study drug to the date of the first observed disease progression (radiological or clinical) or death due to any cause, if death occurred before progression was documented. PFS for participants without tumor progression at the time of analysis was censored at their last date of tumor evaluation.
Time Frame: Up to 2 years
Population: as for outcome 28
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rogaratinib Total Dose Escalation | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 21 | 22 | 70 | 7 | 37
Days | 45 [41 to 88] | 47 [38 to 231] | 105 [80 to 109] | 44 [24 to 144] | 84 [50 to 100]

30. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from start of study treatment until first observed disease progression (radiological or clinical). Progression is defined using RECIST v1.0, as at least a 20% increase in the sum of diameters of the target lesions, taking as a references the smallest sum on study.
Time Frame: Up to 2 years
Population: as for outcome 28
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rogaratinib Total Dose Escalation | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 21 | 22 | 70 | 7 | 37
Days | 45 [41 to 76] | 47 [38 to 231] | 105 [80 to 109] | 68 [35 to 295] | 85 [50 to 105]

31. Secondary Outcome: Duration of Response (DOR)
Description: DOR (for partial and complete response (PR/CR)) was defined as the time (days) from the first documented objective response of PR or CR, whichever was noted earlier, to disease progression or death (if death occurred before progression was documented). DOR was calculated for responders only, i.e. participants with complete or partial response. Therefore, the dose escalation group is not displayed.
Time Frame: Up to 2 years
Population: Participants with a documented objective response of PR or CR.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 1 | 15 | 1 | 2
Days | 522 [NA to NA] — Not Calculated | 126 [63 to 464] | 105 [NA to NA] — Not Calculated | 225 [65 to 385]

32. Secondary Outcome: Duration of Treatment (DOT)
Time Frame: Up to 2 years
Population: as for outcome 28
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rogaratinib Total Dose Escalation | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 21 | 22 | 70 | 7 | 37
Days | 51 [39 to 80] | 82 [43 to 126] | 106 [86 to 119] | 49 [12 to 147] | 84 [51 to 119]

33. Secondary Outcome: Evaluation of Biomarker Status -Change in Serum FGF23 (Fibroblast Growth Factor 23) Levels From Baseline to C2D1
Description: Change in serum FGF23 levels from baseline to C2D1 was reported as ratio to baseline (%).
Time Frame: From baseline to C2D1
Population: All participants with FGF23 data available, and participants from expansion groups were combined as pre-specified in the Statistical Analysis Plan.
Measure: Mean (Standard Deviation); unit: Ratio to baseline (%)
Groups:
- Rogaratinib 800 mg BID: Participants received Rogaratinib as a single dose of 800 mg tablet on C1D1 and 800 mg tablet BID (in total 1600 mg) from C1D3 ongoing in a 21-days Cycle in dose escalation phase.
- Rogaratinib Dose Expansion: All participants from MTD expansion cohorts.
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib Dose Expansion
Number analyzed (Participants) | 2 | 1 | 2 | 2 | 3 | 4 | 48
Ratio to baseline (%) | 201.5 (106.3) | 149.9 | 441.9 (346.2) | 528.0 (290.4) | 402.2 (35.2) | 517.7 (261.0) | 487.0 (447.7)

34. Secondary Outcome: Evaluation of Pharmacodynamic Parameters (PD) - Change of Heart Rate (HR) From Baseline to End of Study
Time Frame: From baseline up to 2 years
Population: Participants received at least one dose of Rogaratinib and have valid data for this outcome measure. Participants were grouped as described in the SAP to allow a comparison of all dose escalation patients (all dose levels pooled together), dose expansion patients (four groups) and total number of patients (overview summaries) in the same table.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Rogaratinib Total Dose Escalation | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 18 | 17 | 62 | 6 | 33
beats per minute | 8.22 (12.47) | 6.41 (15.60) | 6.40 (14.40) | 1.42 (11.65) | 6.27 (15.02)

35. Secondary Outcome: Evaluation of Pharmacodynamic Parameters (PD) - Change of Blood Pressure (BP) From Baseline to End of Study
Time Frame: From baseline up to 2 years
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rogaratinib Total Dose Escalation | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 18 | 17 | 62 | 6 | 33
mmHg
  Systolic Blood Pressure | -1.33 (16.44) | -4.65 (16.73) | -2.56 (19.45) | -5.00 (12.37) | -1.83 (18.85)
  Diastolic Blood Pressure | -2.50 (13.50) | -4.76 (6.99) | -0.63 (12.08) | -0.58 (9.23) | 0.41 (12.55)

36. Secondary Outcome: Evaluation of Pharmacodynamic Parameters (PD) - Change of QT Intervals From Baseline up to Cycle 1, Day 15
Time Frame: From baseline up to Cycle 1, Day 15
Population: Safety Analysis Set (SAF): All participants who received at least one dose of the study medication, and valid data for this outcome measure, and participants from dose escalation groups were combined as pre-specified in the Statistical Analysis Plan.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Rogaratinib Total Dose Escalation | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 21 | 22 | 19 | 6 | 18
msec | 0.60 (23.11) | 12.86 (24.16) | 7.82 (29.39) | 2.89 (16.47) | 6.41 (21.14)

37. Secondary Outcome: Evaluation of Relative Bioavailability of the Tablet Formulation in Comparison to the Solution Formulation of BAY1163877
Description: In order to evaluate the relative bioavailability of the tablet formulation, tablet Cmax/D, AUC(0-tlast)/D, and AUC/D on Cycle 1, Day -3 were compared to solution Cmax/D, AUC(0-tlast)/D, AUC/D on Cycle 1, Day 1 for all analytes. The logarithms of the PK parameters were analyzed using analysis of variance (ANOVA) including participant and formulation effects. Based on these analyses, point estimates (LS-means) and exploratory 90% confidence intervals for the ratios (tablet/solution) of Cmax/D, AUC(0- tlast)/D, and AUC/D were calculated by re-transformation of the logarithmic data using the intra-individual standard deviation of the ANOVA.
Time Frame: On Cycle 1, Day -3 and Cycle 1, Day 1
Population: Only participants who received both tablet and solution formulation were included in the analysis.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Rogaratinib 100 mg BID
Number analyzed (Participants) | 4
ratio
  AUC(0-tlast)/D | 0.9945 [0.7698 to 1.2847]
  AUC/D | 0.9776 [0.7609 to 1.2561]
  Cmax/D | 0.6335 [0.4343 to 0.9240]

38. Secondary Outcome: Tmax (Time to Reach Maximum Drug Concentration in Plasma) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3 and Cycle 1, Day 1
Description: Tmax (time to reach maximum drug concentration in plasma) of BAY1163877 after single dose administration on Cycle 1, Day -3 and Cycle 1, Day 1. Median and full range were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hour(s) post-dose
Population: All participants with valid PK data on Cycle 1, Day -3 and on Cycle 1, Day 1. Some of the participants from the expansion cohorts were included in Rogaratinib expansion food effect, and participants who received 800 mg BID in either escalation or expansion phase were combined as pre-specified in the Statistical Analysis Plan.
Measure: Median (Full Range); unit: hours
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 4 | 3 | 4 | 4 | 51 | 11 | 19 | 13 | 2 | 13
hours
  Cycle 1, Day -3: number analyzed (Participants) | 3 | 4 | 4 | 3 | 4 | 4 | 51 | 10 | 19 | 13 | 2 | 13
  Cycle 1, Day -3 | NA [NA to NA] — No data at the time point | 2.02 [0.983 to 3.03] | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | 2.99 [1.00 to 6.00] | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point
  Cycle 1, Day 1 | 0.633 [0.550 to 0.983] | 0.783 [0.533 to 0.983] | 1.02 [0.617 to 3.25] | 1.02 [1.00 to 1.08] | 1.54 [1.08 to 2.07] | 2.53 [0.517 to 4.05] | 2.00 [0.483 to 4.05] | 2.00 [0.517 to 8.00] | 2.00 [0.500 to 3.25] | 1.00 [0.483 to 2.00] | 1.28 [0.517 to 2.05] | 2.02 [0.500 to 4.00]

39. Secondary Outcome: Tlast (Time of Last Plasma Concentration Above LLOQ) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3 and Cycle 1, Day 1
Description: Tlast (time of last plasma concentration above LLOQ) of BAY1163877 after single dose administration on Cycle 1, Day -3 and Cycle 1, Day 1. Median and full range were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hour(s) post-dose
Population: as for outcome 38
Measure: Median (Full Range); unit: hours
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 4 | 3 | 4 | 4 | 51 | 11 | 19 | 13 | 2 | 13
hours
  Cycle 1, Day -3: number analyzed (Participants) | 3 | 4 | 4 | 3 | 4 | 4 | 51 | 10 | 19 | 13 | 2 | 13
  Cycle 1, Day -3 | NA [NA to NA] — No data at the time point | 48.1 [47.9 to 48.4] | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | 48.0 [46.6 to 48.3] | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point | NA [NA to NA] — No data at the time point
  Cycle 1, Day 1 | 47.7 [46.4 to 47.8] | 47.9 [23.9 to 48.3] | 47.9 [6.0 to 48.6] | 46.9 [24.1 to 48.0] | 48.0 [47.7 to 48.1] | 47.9 [47.8 to 49.5] | 47.9 [11.6 to 49.5] | 47.6 [8.0 to 48.2] | 47.9 [45.9 to 48.5] | 48.0 [11.6 to 49.5] | 48.2 [48.1 to 48.3] | 47.8 [12.0 to 48.7]

40. Secondary Outcome: T1/2 (Half-life Associated With the Terminal Slope) of BAY1163877 After Single Dose Administration on Cycle 1, Day -3 and Cycle 1, Day 1
Description: T1/2 (half-life associated with the terminal slope) of BAY1163877 after single dose administration on Cycle 1, Day -3 and Cycle 1, Day 1. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hour(s) post-dose
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 4 | 3 | 46 | 10 | 18 | 11 | 2 | 12
hours
  Cycle 1, Day -3 | NA (NA) — No data at the time point | 8.15 (22.3) | NA (NA) — No data at the time point | NA (NA) — No data at the time point | NA (NA) — No data at the time point | NA (NA) — No data at the time point | NA (NA) — No data at the time point | 8.22 (31.6) | NA (NA) — No data at the time point | NA (NA) — No data at the time point | NA (NA) — No data at the time point | NA (NA) — No data at the time point
  Cycle 1, Day 1 | 8.34 (24.9) | 8.93 (40.2) | 7.51 (19.2) | 7.93 (54.2) | 8.51 (29.4) | 9.29 (9.86) | 11.7 (44.3) | 12.5 (38.7) | 12.3 (52.1) | 11.5 (42.7) | 14.1 (57.7) | 11.4 (41.0)

41. Secondary Outcome: Tmax,md (Time to Reach Maximum Drug Concentration in Plasma After Multiple-dose Administration) of BAY1163877 on Cycle 1, Day 15
Description: Tmax,md (time to reach maximum drug concentration in plasma after multiple-dose administration) of BAY1163877. Median and full range were reported.
Time Frame: pre-dose (before morning dose), and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
Population: as for outcome 19
Measure: Median (Full Range); unit: hours
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 4 | 70 | 7 | 15 | 27 | 1 | 23
hours | 0.80 [0.50 to 1.10] | 1.08 [0.50 to 1.13] | 1.12 [1.05 to 4.02] | 2.08 [0.50 to 2.17] | 2.10 [2.00 to 3.08] | 2.56 [1.05 to 5.53] | 2.00 [0.00 to 5.53] | 3.17 [1.00 to 4.03] | 1.98 [0.500 to 4.00] | 1.98 [0.500 to 4.07] | 2.07 [2.07 to 2.07] | 2.00 [0.000 to 4.00]

42. Secondary Outcome: Tlast,md (Time of Last Plasma Concentration Above LLOQ After Multiple-dose Administration) of BAY1163877 on Cycle 1, Day 15
Description: Tlast,md (time of last plasma concentration above LLOQ after multiple-dose administration) of BAY1163877. Median and full range were reported.
Time Frame: pre-dose (before morning dose), and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
Population: as for outcome 19
Measure: Median (Full Range); unit: hours
Arm/Group | Rogaratinib 50 mg BID | Rogaratinib 100 mg BID | Rogaratinib 200 mg BID | Rogaratinib 400 mg BID | Rogaratinib 600 mg BID | Rogaratinib 800 mg BID | Rogaratinib 800 mg BID Pooled | Rogaratinib Expansion Food Effect | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 4 | 70 | 7 | 15 | 27 | 1 | 23
hours | 9.80 [6.08 to 11.8] | 11.7 [11.6 to 12.3] | 11.6 [8.00 to 12.6] | 11.7 [11.5 to 11.7] | 11.6 [11.5 to 11.8] | 11.7 [11.1 to 12.0] | 11.7 [6.00 to 12.4] | 11.7 [8.62 to 12.1] | 11.5 [7.83 to 12.0] | 12.0 [8.40 to 12.4] | 11.4 [11.4 to 11.4] | 11.7 [6.00 to 12.0]

ADVERSE EVENTS:
Time Frame: From the first study drug administration up to 30 days after the end of treatment with study drug.
Description: The safety data were reported in groups as pre-specified in the Statistical Analysis Plan, and participants in the Dose Escalation phase were combined.
Groups:
- Rogaratinib Dose Expansion (All Comers): Subjects with cancer types other than bladder cancer (BC), squamous cell carcinoma of the head and neck (SCCHN), and squamous non-small cell lung cancer (sqNSCLC) received 800 mg Rogaratinib oral tablet BID (1600 mg/day) in 21-days cycles.
- Rogaratinib Dose Expansion (BC): Subjects with bladder cancer (BC) received 800 mg Rogaratinib oral tablet BID (1600 mg/day) in 21-days cycles.
- Rogaratinib Dose Expansion (SCCHN): Subjects with squamous cell carcinoma of the head and neck (SCCHN) received 800 mg Rogaratinib oral tablet BID (1600 mg/day) in 21-days cycles.
- Rogaratinib Dose Expansion (sqNSCLC): Subjects with squamous non-small cell lung cancer (sqNSCLC) received 800 mg Rogaratinib oral tablet BID (1600 mg/day) in 21-days cycles.
Arm/Group | Rogaratinib Total Dose Escalation | Rogaratinib Dose Expansion (All Comers) | Rogaratinib Dose Expansion (BC) | Rogaratinib Dose Expansion (SCCHN) | Rogaratinib Dose Expansion (sqNSCLC)
All-Cause Mortality (participants affected / at risk) | 3/23 | 6/23 | 17/74 | 2/8 | 12/40
Serious Adverse Events (participants affected / at risk) | 9/23 | 14/23 | 44/74 | 5/8 | 24/40
Other Adverse Events (participants affected / at risk) | 22/23 | 23/23 | 73/74 | 8/8 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rogaratinib Total Dose Escalation (N=23) | Rogaratinib Dose Expansion (All Comers) (N=23) | Rogaratinib Dose Expansion (BC) (N=74) | Rogaratinib Dose Expansion (SCCHN) (N=8) | Rogaratinib Dose Expansion (sqNSCLC) (N=40)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 5 (7) | 1 (2) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (2) | 2 (3) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (5) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dural arteriovenous fistula (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (4)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 5 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rogaratinib Total Dose Escalation (N=23) | Rogaratinib Dose Expansion (All Comers) (N=23) | Rogaratinib Dose Expansion (BC) (N=74) | Rogaratinib Dose Expansion (SCCHN) (N=8) | Rogaratinib Dose Expansion (sqNSCLC) (N=40)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (11) | 17 (29) | 3 (6) | 12 (19)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (3) | 12 (13) | 1 (2) | 3 (3)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (2)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Growth of eyelashes (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pingueculitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 11 (14) | 0 (0) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 10 (16) | 25 (41) | 3 (4) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 4 (8) | 13 (20) | 48 (106) | 4 (5) | 23 (42)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 25 (42) | 0 (0) | 9 (13)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (3) | 5 (5) | 1 (1) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 8 (11) | 20 (31) | 4 (4) | 11 (19)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (3) | 11 (18) | 1 (2) | 8 (13)
Vomiting (Gastrointestinal disorders) | 2 (4) | 1 (1) | 13 (18) | 2 (3) | 6 (7)
Asthenia (General disorders) | 0 (0) | 3 (8) | 14 (35) | 2 (3) | 5 (10)
Chest pain (General disorders) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 5 (6)
Fatigue (General disorders) | 7 (8) | 7 (12) | 28 (55) | 2 (3) | 11 (22)
Mucosal inflammation (General disorders) | 0 (0) | 1 (4) | 4 (7) | 0 (0) | 1 (1)
Oedema (General disorders) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (5) | 4 (5) | 1 (2) | 4 (6)
Pyrexia (General disorders) | 2 (3) | 6 (8) | 7 (11) | 0 (0) | 6 (8)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 3 (5) | 6 (9) | 0 (0) | 3 (4)
Pneumonia (Infections and infestations) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 7 (10)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 5 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 19 (32) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 4 (5) | 8 (20) | 0 (0) | 8 (12)
Amylase increased (Investigations) | 0 (0) | 2 (4) | 6 (20) | 0 (0) | 5 (14)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 5 (6) | 9 (19) | 0 (0) | 9 (14)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (5) | 7 (9) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 4 (7) | 1 (7) | 3 (4)
Blood creatinine increased (Investigations) | 0 (0) | 3 (4) | 12 (24) | 2 (3) | 6 (11)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 7 (16) | 0 (0) | 3 (4)
Lipase increased (Investigations) | 1 (1) | 3 (13) | 10 (40) | 1 (5) | 10 (25)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 5 (7) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 4 (7)
Blood phosphorus increased (Investigations) | 11 (21) | 20 (58) | 31 (88) | 5 (11) | 31 (85)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 7 (12) | 1 (1) | 3 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 5 (13) | 7 (10) | 0 (0) | 8 (18)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 3 (5)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 6 (11) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (25) | 1 (4) | 4 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (6) | 2 (3) | 4 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 6 (10) | 0 (0) | 1 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 5 (6) | 0 (0) | 3 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 2 (4)
Decreased appetite (Metabolism and nutrition disorders) | 5 (9) | 10 (12) | 29 (50) | 4 (9) | 16 (18)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 5 (9) | 17 (30) | 1 (1) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 12 (17) | 0 (0) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 8 (8) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 6 (9) | 1 (3) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 3 (4)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 5 (7) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 4 (5) | 0 (0) | 7 (7)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (3) | 17 (20) | 2 (3) | 7 (8)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (6) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (5) | 3 (3) | 2 (2) | 4 (5)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 9 (13) | 0 (0) | 2 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 4 (4) | 7 (8) | 0 (0) | 13 (20)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 6 (9) | 0 (0) | 12 (20)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 4 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (10) | 0 (0) | 7 (7)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 3 (5)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 6 (6) | 20 (23) | 0 (0) | 8 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 17 (22) | 2 (2) | 4 (6)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 7 (8) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 7 (13) | 0 (0) | 3 (3)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (7) | 1 (1) | 0 (0) | 0 (0)
Nail hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 12 (22) | 1 (2) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 7 (16) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 3 (6)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 3 (9)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (2) | 1 (2) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT01976741/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT01976741/SAP_001.pdf